CLINICAL TRIAL: NCT00030498
Title: Phase I Study of OSI-774 (NSC 718781) for Solid Tumors in Patients With Hepatic or Renal Dysfunction
Brief Title: Erlotinib in Treating Patients With Solid Tumors and Liver or Kidney Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01868; CALGB-60101; U10CA031946 (NIH); CDR0000069170 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Ependymoma; Adult Anaplastic Oligodendroglioma; Adult Brain Stem Glioma; Adult Diffuse Astrocytoma; Adult Ependymoblastoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Adult Myxopapillary Ependymoma; Adult Oligodendroglioma; Adult Pilocytic Astrocytoma; Adult Primary Hepatocellular Carcinoma; Adult Subependymoma; Advanced Adult Primary Liver Cancer; Advanced Malignant Mesothelioma; Male Breast Cancer; Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Adult Brain Tumor; Recurrent Adult Primary Liver Cancer; Recurrent Anal Cancer; Recurrent Basal Cell Carcinoma of the Lip; Recurrent Bladder Cancer; Recurrent Breast Cancer; Recurrent Cervical Cancer; Recurrent Colon Cancer; Recurrent Esophageal Cancer; Recurrent Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Recurrent Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Lymphoepithelioma of the Oropharynx; Recurrent Malignant Mesothelioma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Non-small Cell Lung Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Pancreatic Cancer; Recurrent Prostate Cancer; Recurrent Rectal Cancer; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage II Esophageal Cancer; Stage II Pancreatic Cancer; Stage III Esophageal Cancer; Stage III Pancreatic Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Adenoid Cystic Carcinoma of the Oral Cavity; Stage IV Anal Cancer; Stage IV Basal Cell Carcinoma of the Lip; Stage IV Bladder Cancer; Stage IV Breast Cancer; Stage IV Colon Cancer; Stage IV Esophageal Cancer; Stage IV Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage IV Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage IV Lymphoepithelioma of the Nasopharynx; Stage IV Lymphoepithelioma of the Oropharynx; Stage IV Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage IV Mucoepidermoid Carcinoma of the Oral Cavity; Stage IV Non-small Cell Lung Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Pancreatic Cancer; Stage IV Prostate Cancer; Stage IV Rectal Cancer; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity; Stage IVA Cervical Cancer; Stage IVB Cervical Cancer; Unspecified Adult Solid Tumor, Protocol Specific; Untreated Metastatic Squamous Neck Cancer With Occult Primary
MeSH Terms: conditions — Astrocytoma; Ependymoma; Oligodendroglioma; Neuroectodermal Tumors, Primitive; Glioblastoma; Gliosarcoma; Glioma; Carcinoma, Hepatocellular; Glioma, Subependymal; Breast Neoplasms, Male; Brain Neoplasms; Anus Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Esthesioneuroblastoma, Olfactory; Mesothelioma, Malignant; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Pancreatic Neoplasms; Prostatic Neoplasms; Rectal Neoplasms; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Erlotinib Hydrochloride

ARMS (1):
- Treatment (erlotinib hydrochloride) (Experimental): Patients receive oral erlotinib once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the effectiveness of erlotinib in treating patients who have metastatic or unresectable solid tumors and liver or kidney dysfunction. Biological therapies such as erlotinib may interfere with the growth of tumor cells and slow the growth of the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of erlotinib in patients with solid tumors and hepatic or renal dysfunction.

II. Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to hepatic or renal dysfunction (albumin less than 2.5 g/dL, direct bilirubin less than 1.0 mg/dL, any AST, and creatinine normal vs direct bilirubin 1.0-7.0 mg/dL, any AST, and creatinine normal vs creatinine 2.5-5.0 mg/dL, albumin 2.5 g/dL or greater, AST less than 3 times upper limit of normal, and direct bilirubin less than 1.0 mg/dL).

Patients receive oral erlotinib once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, at least 6 evaluable patients are treated at that dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor, including gliomas and the following epithelial malignancies:

  * Non-small cell lung
  * Mesothelioma
  * Breast
  * Head and neck
  * Esophageal
  * Pancreatic
  * Bladder
  * Prostate
  * Ovarian
  * Anal
  * Colorectal carcinoma
  * Cervical carcinoma
  * Hepatocellular carcinoma
* Metastatic or unresectable disease
* Standard curative or palliative therapy does not exist or is no longer effective
* Epidermal growth factor receptor (EGFR) positive
* Hepatic or renal dysfunction defined as one of the following:

  * Direct bilirubin 1.0-7.0 mg/dL with any AST
  * Albumin less than 2.5 g/dL
  * Creatinine 2.5-5.0 mg/dL
* Brain metastases allowed provided patient is asymptomatic, previously treated, has stable disease for at least 2 months, and is not currently receiving steroid therapy
* Hormone receptor status:

  * Not specified
* Male or female
* Performance status - ECOG 0-2
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* See Disease Characteristics
* No evidence of biliary obstruction
* See Disease Characteristics
* No evidence of renal obstruction
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No gastrointestinal tract disease that would preclude ability to take oral medications
* No requirement for IV alimentation
* No active peptic ulcer disease
* No prior corneal abnormalities (e.g., dry eye syndrome or Sjogren's syndrome)
* No prior congenital abnormality (e.g., Fuch's dystrophy)
* No prior abnormal slit-lamp exam using a vital dye (e.g., fluorescein or Bengal-Rose)
* No prior abnormal corneal sensitivity test (e.g., Schirmer test or similar tear production test)
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)
* At least 4 weeks since prior chemotherapy (6 weeks for melphalan or mitomycin)
* No prior nitrosoureas
* See Disease Characteristics
* No concurrent steroids
* At least 4 weeks since prior radiotherapy
* At least 4 weeks since prior major surgery
* No prior surgical procedures affecting absorption
* No prior EGFR-targeting therapies, including gefitinib or Imclone C-225
* At least 3 months since prior suramin
* More than 7 days since prior grapefruit juice
* More than 7 days since other prior CYP3A4 inhibitors
* No concurrent grapefruit juice
* No concurrent CYP3A4 inducers, substrates, or other inhibitors
* No concurrent medications known to affect hepatic or renal function, including antiseizure medication or nonsteroidal anti-inflammatory agents
* No concurrent combination anti-retroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2001-12; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of OSI-774 determined by dose-limiting toxicities | Within the first 4 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Antonius Miller, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States